CLINICAL TRIAL: NCT06220526
Title: A Prospective Randomized Clinical Trial Comparing Menghini-type Needle and Franseen-type Needle for Endobronchial Ultrasound-guided Transbronchial Needle Aspiration for Pathological Diagnosis of Sarcoidosis
Brief Title: Comparing Menghini-type Needle and Franseen-type Needle in EBUS-TBNA for Sarcoidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kazuhiro Yasufuku, Department Head. Division of Thoracic Surgery, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-5265
Record Dates: First submitted 2023-11-27; First posted 2024-01-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Suspected Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menghini-type needle (Other): the standard needle type
  Interventions: Device: endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA)
- Franseen-type needles (Active Comparator): the active comparator arm
  Interventions: Device: endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA)

INTERVENTIONS:
Device: endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) — Transbronchial biopsy with Menghini-type or Franseen type Needle

SUMMARY:
This randomized pilot clinical trial aims to examine whether sample collection with Franseen-type needles are effective for the diagnosis of sarcoidosis, as defined by improved sample quality for pathological diagnosis compared to the conventional Menghini-type needle.

DETAILED DESCRIPTION:
This study is a prospective randomized control trial. More than 370 lymph nodes from approximately 128 patients with enlarged mediastinal and/or hilar lymph nodes (≥10 mm short-axis diameter on CT scan) and suspected sarcoidosis will be enrolled in this study. This is a single-center study conducted at the Toronto General Hospital.

If consent is obtained, patients will be considered enrolled. The patients will then be assigned to either Menghini-type (the standard needle type in Toronto General Hospital) or Franseen-type needles in a 1:1 ratio with stratified randomization by the availability of rapid on-site cytology evaluation. An automated randomization program will be used to generate the randomization scheme for the study. Samples from mediastinal and hilar lymph nodes will be obtained by EBUS-guided Menghini-type or Franseen-type needle biopsy. Post-procedural assessment will take place in the endoscopy recovery room and will include, but not limited to, monitoring of vital signs, signs of bleeding, and pulmonary status. As EBUS-TBNA is an outpatient procedure, patients will be discharged home after the procedure.

Specimens (cell pellet and/or tissue fragment) will be assessed by pathologists as per their usual practice. The pathologists will remain blinded to the allocated needle. Specimens will be classified by their adequacy for histological assessment and diagnostic yield. In addition, total procedure time and mean number of needle passes to obtain tissue samples will be compared between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* -Any adult patient aged 18 years or older with enlarged mediastinal and/or hilar lymph nodes
* (≥10 mm short-axis diameter on a CT scan), suspected as having sarcoidosis based on clinical
* history, physical exam, and other investigations, and booked for EBUS-TBNA.

Exclusion Criteria:

* -Patients that are unable to provide informed consent

  - Patients with lymphadenopathy strongly suspected to be secondary to other diseases based on
* clinical history, physical exam, and/or other investigations (e.g., lung cancer, lymphoma,
* infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of adequate tissue sampling from lymph nodes (as determined by pathologists) | 3 years
  To compare the performance characteristics of endobronchial ultrasound-guided transbronchial needle aspiration with Menghini-type needle and Franseen-type needle

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No